CLINICAL TRIAL: NCT02875249
Title: Chemotherapy-driven Dysbiosis in the Intestinal Microbiome
Brief Title: Intestinal Microbiome and Chemotherapy
Acronym: EMAAD
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/10/04-Q
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Diarrhea
Keywords: post-antibiotic diarrhea; intestinal microbiome
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool of patients for bacterial analysis
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: patients stool collection — patients stool collection

SUMMARY:
Chemotherapy is commonly used as myeloablative conditioning treatment to prepare patients for haematopoietic stem cell transplantation (HSCT). Chemotherapy leads to several side effects, with gastrointestinal (GI) mucositis being one of the most frequent. Current models of GI mucositis pathophysiology are generally silent on the role of the intestinal microbiome.

The aim of the study is to identify functional mechanisms by which the intestinal microbiome may play a key role in the pathophysiology of GI mucositis, the investigators applied high throughput DNA-sequencing analysis to identify microbes and microbial functions that are modulated following chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-Hodgkin's lymphoma
* Participants receiving the same myeloablative conditioning regimen for five consecutive days, including high-dose Carmustine (Bis-chloroethylnitrosourea), Etoposide, Aracytine and Melphalan.

Exclusion Criteria:

* Patients with a history of Inflammatory Bowel Diseases (IBD), exposed to probiotics, prebiotics or broad-spectrum antibiotics, or administered nasal-tube feeding or parenteral nutrition in the month prior to initiation of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, men and women, 18 to 65, who receive intravenous antibiotics broad spectrum (Tazocilline (piperacillin tazobactam) and Amiklin (amikacin)) in support of the context of febrile neutropenia following a autologous stem cells.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
analyze of the fecal samples using 16S ribosomal ribonucleic acid (rRNA) gene sequencing | baseline
analyze of the fecal samples using 16S ribosomal ribonucleic acid (rRNA) gene sequencing | at day 7

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Montassier, PH, Principal Investigator — Nantes Univetsity Hospital

IPD SHARING:
Plan to Share IPD: No